CLINICAL TRIAL: NCT04118257
Title: Effects of Short-term Sugary Beverage Consumption on Type-2 Diabetes and Cardiovascular Disease Risk Factors: A Randomized Controlled Trial
Brief Title: Short-term Sugary Beverage Consumption on Glucose Control and Cardiovascular Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Sara K Rosenkranz, Principal Investigator, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro8531
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Metabolic Syndrome
Keywords: Glucose control; Cardiovascular disease risk factors; Sugary beverages; Pulmonary function
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruit Juice (Experimental): Participants consumed 2 bottles of 100% fruit juice daily for 3 weeks.
  Interventions: Dietary Supplement: Sugary beverage: Fruit juice
- Soda (Experimental): Participants consumed 2 cans of caffeine-free Coca Cola daily for 3 weeks.
  Interventions: Dietary Supplement: Sugary beverage: Soda
- Water (Other): Participants consumed 2 bottles of water daily for 3 weeks.
  Interventions: Dietary Supplement: Control: Water

INTERVENTIONS:
Dietary Supplement: Sugary beverage: Fruit juice — Participants consumed 100% fruit juice (~710mL) daily for three weeks, along with their habitual diets.
  Arms: Fruit Juice
Dietary Supplement: Sugary beverage: Soda — Participants consumed soda (~710mL) daily for three weeks, along with their habitual diets.
  Arms: Soda
Dietary Supplement: Control: Water — Participants consumed water (~710mL) daily for three weeks, along with their habitual diets.
  Arms: Water

SUMMARY:
Our goal is to determine how the addition of sugar-sweetened beverages to the diet affects glucose control, cardiovascular disease risk factors, and pulmonary function in healthy, young adults.

DETAILED DESCRIPTION:
In a 3-arm randomized controlled trial, 36 participants consumed one of three beverages for three weeks: water (W), caffeine-free soda (S), or 100% fruit juice (FJ). Participants consumed two servings/day (~710mL) of their randomized beverage for three weeks, along with their habitual diets. At baseline and following the 3-week intervention, participants completed glucose control, cardiovascular disease risk factor, and pulmonary function assessments.

ELIGIBILITY:
Inclusion Criteria:

* Free from diagnosis of diabetes and pulmonary illness
* Have no intake of glucose or lipid lowering medication.

Exclusion Criteria:

* Smoke
* Currently pregnant
* Have bronchitis
* Have more than 2 risk factors for cardiovascular disease, as defined by the American College of Sports Medicine (ACSM).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Change in glucose iAUC | Week 0 and Week 3
  Glucose obtained from blood sample in a fasted state and in response to a meal

SECONDARY OUTCOMES:
Change in plasma lipids | Week 0 and Week 3
  Total cholesterol (TC), LDL-c , VLDL-c, HDL-c , triglycerides (TG) from blood sample in a fasted state and following consumption of a meal
Change in homeostatic model assessment for insulin resistance | Week 0 and Week 3
  Calculated from fasting glucose and insulin values
Change in blood pressure | Week 0 and Week 3
  Evaluated via automated sphygmomanometer.
Change in BMI | Week 0 and Week 3
  Weight and height will be combined to report BMI in kg/m^2
Change in pulmonary function | Week 0 and Week 3
  Assessed using the maximum flow-volume loop
Change in insulin iAUC | Week 0 and Week 3
  Glucose obtained from blood sample in a fasted state and in response to a meal
Change in serum fructosamine | Week 0 and Week 3
  Fructosamine obtained from blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rosenkranz, PhD, Principal Investigator — Kansas State University
Locations (1):
- Lafene Health Center, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No